CLINICAL TRIAL: NCT05794893
Title: Good Behavior Game - a Randomized Controlled Study Among Young Children in Swedish Primary Schools.
Brief Title: Effects of Good Behavior Game in a Swedish Sample
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-06804
Record Dates: First submitted 2023-03-08; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Problem Behavior
Keywords: Problem Behavior; School; Prevention
MeSH Terms: conditions — Problem Behavior

STUDY DESIGN:
Intervention Model Description: All participants in the intervention group receive the same GBG intervention. The control condition consists of service-as-usual (SAU).
Who Masked: Outcomes Assessor
Masking Description: The independent assessors are blind to conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Good Behavior Game (Experimental): 28 classes receiving Good Behavior Game intervention
  Interventions: Behavioral: Good Behavior Game
- Service-as-usual (No Intervention): 16 classes receiving usual classroom teaching

INTERVENTIONS:
Behavioral: Good Behavior Game — Universal school-based intervention reinforcing prosocial behaviors and discouraging disruptive behaviors in young students.
  Arms: Good Behavior Game

SUMMARY:
This project seeks to study the impact of Good Behavior Game (GBG), a behavior management program, on classroom environment and problem behavior in K-3 classrooms.

The goal of this randomized trial is to study the impact of Good Behavior Game (GBG), a behavior management program, on classroom environment and problem behavior in K-3 classrooms in Sweden. The main question it aims to answer is:

• Does GBG decrease problem behaviors in K-3 classrooms?

Teachers in the intervention group will be trained in GBG and asked to implement it in their respective classrooms. Teachers in the comparison group will provide usual practice.

DETAILED DESCRIPTION:
Background: Early conduct problems are prevalent and a prominent risk factor for several adverse health-related and psychosocial outcomes in later life. Good Behavior Game (GBG) is a promising school-based behavior management program with the potential of reaching many children in their formative years.

Primary objective: To study the effectiveness of Good Behavior Game in reducing problem behaviors in Swedish K-3 classrooms under real-world conditions.

Secondary objectives: To investigate changes in problem behaviors in common school areas, classroom climate, teacher collective efficacy, on-task behavior, and behavioral management practices as a result of teacher training in GBG. The study also seeks to investigate implementation as a moderator, as well as potential barriers and facilitators in regards to implementation.

Type of trial: Cluster-randomized controlled trial

Trial design and methods: Recruitment of schools in a Swedish municipality started early 2021. In May 2021, 5 schools were randomized to either intervention group or wait-list (service-as-usual). Data collection started in August 2021 and ended in June 2022. The intervention group received training in GBG from September 2021 to May 2022 by certified trainers who also collected fidelity data through observations throughout the school year. Teacher ratings and observer data was collected at baseline (August 2021), along with a first (November 2021) and second follow-up (May 2022, primary endpoint) throughout the first school year of implementation.

Statistical methodology and analysis: Statistical analysis will primarily include frequentist intent-to-treat analysis, and comparisons of estimates with a corresponding Bayesian model using weakly informative priors.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility is based on school or classroom level factors. Schools must have at least one classroom with a group of students enrolled in grades K, 1, 2, or 3.

Exclusion Criteria:

* Special education classrooms are not eligible, though inclusive classrooms with a minority of students needing special education can be included.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
Teacher-rated problem behavior in the classroom | Baseline
  A teacher-rated scale listing 20 common problem behaviors in the classroom. The teachers bases their ratings on the week before. Every item is rated on a scale from 0 (no times last week) to 4 (several times a day).
Teacher-rated problem behavior in the classroom | 3 months
  A teacher-rated scale listing 20 common problem behaviors in the classroom. The teachers bases their ratings on the week before. Every item is rated on a scale from 0 (no times last week) to 4 (several times a day).
Teacher-rated problem behavior in the classroom | 9 months (primary endpoint)
  A teacher-rated scale listing 20 common problem behaviors in the classroom. The teachers bases their ratings on the week before. Every item is rated on a scale from 0 (no times last week) to 4 (several times a day).

SECONDARY OUTCOMES:
Classroom Atmosphere Measure | Baseline
  Measure of 10 different behavioral classroom factors rated by an independent observer after 30 minutes of observing a classroom. The observer scores every item on a scale from 1-5, were 1 is generally considered very low and 5 is considered very high. A rating of 0 is used when the item/factor is not applicable or possible to rate. The following items are rated:
  1. Students' level of compliance during structured time
  2. Students seem to handle transitions well
  3. Students consistently follow rules appropriate to settings
  4. Students' level of cooperation
  5. Students attempt problem-solving
  6. Students express feelings appropriately
  7. Students' level of interest/enthusiasm/involvement
  8. Classroom is focused and on-task
  9. Classroom responsive to individual differences in students' needs, feelings, etc.
  10. Classroom is supportive of students' efforts
Classroom Atmosphere Measure | 3 months
  Measure of 10 different behavioral classroom factors rated by an independent observer after 30 minutes of observing a classroom. The observer scores every item on a scale from 1-5, were 1 is generally considered very low and 5 is considered very high. A rating of 0 is used when the item/factor is not applicable or possible to rate. The following items are rated:
  1. Students' level of compliance during structured time
  2. Students seem to handle transitions well
  3. Students consistently follow rules appropriate to settings
  4. Students' level of cooperation
  5. Students attempt problem-solving
  6. Students express feelings appropriately
  7. Students' level of interest/enthusiasm/involvement
  8. Classroom is focused and on-task
  9. Classroom responsive to individual differences in students' needs, feelings, etc.
  10. Classroom is supportive of students' efforts
Classroom Atmosphere Measure | 9 months
  Measure of 10 different behavioral classroom factors rated by an independent observer after 30 minutes of observing a classroom. The observer scores every item on a scale from 1-5, were 1 is generally considered very low and 5 is considered very high. A rating of 0 is used when the item/factor is not applicable or possible to rate. The following items are rated:
  1. Students' level of compliance during structured time
  2. Students seem to handle transitions well
  3. Students consistently follow rules appropriate to settings
  4. Students' level of cooperation
  5. Students attempt problem-solving
  6. Students express feelings appropriately
  7. Students' level of interest/enthusiasm/involvement
  8. Classroom is focused and on-task
  9. Classroom responsive to individual differences in students' needs, feelings, etc.
  10. Classroom is supportive of students' efforts
Classroom Environment Scale | Baseline
  Teacher rates 15 items about the classroom climate (e.g. how well students cooperate, task-orientation etc.). The items are rated on a 0-3 likert scale, some being reverse-coded.
Classroom Environment Scale | 9 months
  Teacher rates 15 items about the classroom climate (e.g. how well students cooperate, task-orientation etc.). The items are rated on a 0-3 likert scale, some being reverse-coded.
On-task behavior: Planned activity check/PLACHECK | Baseline
  Group-based measure of on task behavior in classroom. Rated by an independent assessor. Score is based on number of children on-task divided by total number of children in the classroom. On-task behavior is rated after 3-minute intervals for a total of 18 minutes. An average of the percentage scores is used as an outcome.
On-task behavior: Planned activity check/PLACHECK | 3 months
  Group-based measure of on task behavior in classroom. Rated by an independent assessor. Score is based on number of children on-task divided by total number of children in the classroom. On-task behavior is rated after 3-minute intervals for a total of 18 minutes. An average of the percentage scores is used as an outcome.
On-task behavior: Planned activity check/PLACHECK | 9 months
  Group-based measure of on task behavior in classroom. Rated by an independent assessor. Score is based on number of children on-task divided by total number of children in the classroom. On-task behavior is rated after 3-minute intervals for a total of 18 minutes. An average of the percentage scores is used as an outcome.
Teacher-rated problem behavior in school | Baseline
  A teacher-rated scale listing 20 common problem behaviors in the school's common/shared areas. The teachers bases their ratings on the week before. Every item is rated on a scale from 0 (no times last week) to 4 (several times a day).
Teacher-rated problem behavior in school | 3 months
  A teacher-rated scale listing 20 common problem behaviors in the school's common/shared areas. The teachers bases their ratings on the week before. Every item is rated on a scale from 0 (no times last week) to 4 (several times a day).
Teacher-rated problem behavior in school | 9 months
  A teacher-rated scale listing 20 common problem behaviors in the school's common/shared areas. The teachers bases their ratings on the week before. Every item is rated on a scale from 0 (no times last week) to 4 (several times a day).
Collective teacher efficacy | Baseline
  Teacher rates 12 items on the perceived efficacy of teachers as a collective being able to teach the students attending the school. Items are rated on a 0-5 likert scale, some being reverse-coded.
Collective teacher efficacy | 9 months
  Teacher rates 12 items on the perceived efficacy of teachers as a collective being able to teach the students attending the school. Items are rated on a 0-5 likert scale, some being reverse-coded.
Positive behavior support | Baseline
  The teacher rates 9 items on their own use of several practices that aim to increase desirable behaviors in the classroom. The teacher will report based on the last 30 days. The items can be rated on a scale from 0 (0 times) to 7 (more than 20 times).
Positive behavior support | 9 months
  The teacher rates 9 items on their own use of several practices that aim to increase desirable behaviors in the classroom. The teacher will report based on the last 30 days. The items can be rated on a scale from 0 (0 times) to 7 (more than 20 times).
Behavioral correction | Baseline
  The teacher rates 8 items on their own use of several practices that aim to punish, reduce or correct undesirable behaviors in the classroom. The teacher will report based on the last 30 days. The items can be rated on a scale from 0 (0 times) to 7 (more than 20 times).
Behavioral correction | 9 months
  The teacher rates 8 items on their own use of several practices that aim to punish, reduce or correct undesirable behaviors in the classroom. The teacher will report based on the last 30 days. The items can be rated on a scale from 0 (0 times) to 7 (more than 20 times).
Observed general praise | Baseline
  An independent observer counts the number of times the teacher uses general praise towards one or more students by the teacher. General praise counts as praise were the behavior eliciting praise is not specified, for example "good job". Can also be non-verbal. The observation and counting lasts for 30 minutes.
Observed general praise | 3 months
  An independent observer counts the number of times the teacher uses general praise towards one or more students by the teacher. General praise counts as praise were the behavior eliciting praise is not specified, for example "good job". Can also be non-verbal. The observation and counting lasts for 30 minutes.
Observed general praise | 9 months
  An independent observer counts the number of times the teacher uses general praise towards one or more students by the teacher. General praise counts as praise were the behavior eliciting praise is not specified, for example "good job". Can also be non-verbal. The observation and counting lasts for 30 minutes.
Observed specific praise | Baseline
  An independent observer counts the number of times behavioral specific praise is used towards one or more students by the teacher. Behavioral specific praise counts as praise or feedback that also entails a description of the behavior eliciting praise, such as "good work reading that out loud". The observation and counting lasts for 30 minutes.
Observed specific praise | 3 months
  An independent observer counts the number of times behavioral specific praise is used towards one or more students by the teacher. Behavioral specific praise counts as praise or feedback that also entails a description of the behavior eliciting praise, such as "good work reading that out loud". The observation and counting lasts for 30 minutes.
Observed specific praise | 9 months
  An independent observer counts the number of times behavioral specific praise is used towards one or more students by the teacher. Behavioral specific praise counts as praise or feedback that also entails a description of the behavior eliciting praise, such as "good work reading that out loud". The observation and counting lasts for 30 minutes.
Observed reprimands | Baseline
  An independent observer counts the number of times reprimands are used towards one or more students by the teacher. Reprimands are verbal or non-verbal cues were the teacher demands on students ceasing a certain behavior or otherwise point out a behavior that should not be occuring. The observation and counting lasts for 30 minutes.
Observed reprimands | 3 months
  An independent observer counts the number of times reprimands are used towards one or more students by the teacher. Reprimands are verbal or non-verbal cues were the teacher demands on students ceasing a certain behavior or otherwise point out a behavior that should not be occuring. The observation and counting lasts for 30 minutes.
Observed reprimands | 9 months
  An independent observer counts the number of times reprimands are used towards one or more students by the teacher. Reprimands are verbal or non-verbal cues were the teacher demands on students ceasing a certain behavior or otherwise point out a behavior that should not be occuring. The observation and counting lasts for 30 minutes.

OTHER OUTCOMES:
Implementation barriers and facilitators | Baseline
  A teacher rates 14 items drawn from the Consolidated Framework for Implementation Research (CFIR). The instrument itself is called The Barrier Buster Tool. The instrument primarily measures contextual factors that are thought to affect implementation and fidelity of a method being implemented. Every item has two ratings. First rating scores if the statement is a barrier (0), neutral (1) or facilitating factor (2). The second column rates the strength of the factor, i.e., if the factor is considered to have a weak/no effect (0) or strong effect (1). Only measured in the experimental group receiving GBG.
Implementation barriers and facilitators | 3 months
  A teacher rates 14 items drawn from the Consolidated Framework for Implementation Research (CFIR). The instrument itself is called The Barrier Buster Tool. The instrument primarily measures contextual factors that are thought to affect implementation and fidelity of a method being implemented. Every item has two ratings. First rating scores if the statement is a barrier (0), neutral (1) or facilitating factor (2). The second column rates the strength of the factor, i.e., if the factor is considered to have a weak/no effect (0) or strong effect (1). Only measured in the experimental group receiving GBG.
Implementation barriers and facilitators | 9 months
  A teacher rates 14 items drawn from the Consolidated Framework for Implementation Research (CFIR). The instrument itself is called The Barrier Buster Tool. The instrument primarily measures contextual factors that are thought to affect implementation and fidelity of a method being implemented. Every item has two ratings. First rating scores if the statement is a barrier (0), neutral (1) or facilitating factor (2). The second column rates the strength of the factor, i.e., if the factor is considered to have a weak/no effect (0) or strong effect (1). Only measured in the experimental group receiving GBG.
Average fidelity of implementation | Monthly observations from baseline to 9 months
  The trainers responsible for coaching in GBG observes and rates to what extent teachers are following the manual during GBG-sessions. The trainers used standardized observation forms detailing several components of a GBG session, such as setting rules and announcing the time frame. Scores will be based on number of items that the trainer rates as completed, divided by the maximum number of items possible to complete in a session. The average score is then calculated from all sessions.
Certification in GBG | 9 months
  A certification of completing training and performing GBG with fidelity as assessed by trainers. A score of 0 means the teacher has not been certified at the end of the school year. A score of 1 means the teacher has been certified at the end of the school year. The requirements for certification are: participating in all 3 workshops, conducting at least 60 sessions, being observed and receiving feedback at least 9 times with the trainers assessing the sessions as having high enough fidelity.

CONTACTS AND LOCATIONS:
Overall Officials: Björn Hofvander, Principal Investigator — Lund University
Locations (5):
- Sweden (5):
  - Johannesskolan, Malmo
  - Klagshamnsskolan, Malmo
  - Malmö friskola, Malmo
  - Monbijouskolan, Malmo
  - Ängsdals skola, Malmo

IPD SHARING:
Plan to Share IPD: No
The study does not collect individual participant data. Only group/aggregated data is collected. This data may be made available to other researchers unless conflicting with regulations, consent or other aspects of the ethical review.

REFERENCES:
- [Derived] Djamnezhad D, Bergstrom M, Delfin C, Hofvander B. Classroom effects of a preventive behavioral management program: A pragmatic cluster-randomized trial of Good Behavior Game. PLOS Ment Health. 2025 Dec 23;2(12):e0000487. doi: 10.1371/journal.pmen.0000487. eCollection 2025. PMID 41662083
- [Derived] Djamnezhad D, Bergstrom M, Andren P, Hofvander B. Good behavior game - study protocol for a randomized controlled trial of a preventive behavior management program in a Swedish school context. Front Psychiatry. 2023 Oct 5;14:1256714. doi: 10.3389/fpsyt.2023.1256714. eCollection 2023. PMID 37867765